CLINICAL TRIAL: NCT05735457
Title: A Short, Animated Storytelling Video to Increase Knowledge About Sodium Intake as a Major Cardiovascular Risk Factor and to Give Recommendations for a Low-sodium Healthy Diet: an Online, Randomized, Controlled Trial
Brief Title: A Short, Animated Storytelling Video to Increase Knowledge About Sodium Intake as a Cardiovascular Risk Factor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Freiburg (Other)
Collaborators: Stanford University (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, PD Dr. Alexander Supady, Attending Physician, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EduEntertainSodium_23
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Sodium Excess; Cardiovascular Risk Factor; Education Entertainment Intervention; Short, Animated Storytelling
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Arm (Experimental): Participants will be shown a short, animated storytelling (SAS) video on dietary sodium and thereafter be asked to complete a questionnaire to assess knowledge on dietary sodium and behavioral expectation.
  Two weeks later, participants will once again be asked to complete the knowledge and behavioral expectation questionnaire.
  Interventions: Other: A short, animated storytelling video on dietary sodium
- Exposed Control Arm (No Intervention): Participants will be asked to complete a questionnaire to assess knowledge on dietary sodium and behavioral expectation (the same questionnaire as in arm 1, however, without being exposed to the SAS video on dietary sodium before.
  Two weeks later, participants will once again be asked to complete the knowledge and behavioral expectation questionnaire.
- Attention Placebo Control Arm (Placebo Comparator): Participants will be shown a attention placebo control (APC) video, unrelated to the outcomes measured in this trial, before being asked to complete the knowledge and behavioral expectation questionnaire.
  Two weeks later, participants will once again be asked to complete the knowledge and behavioral expectation questionnaire.
  Interventions: Other: A short, animated storytelling attention placebo video
- Un-exposed Control Arm (No Intervention): Participants will not view a video and will not be asked to complete the questionnaire.
  Two weeks later, participants will once again be asked to complete the knowledge and behavioral expectation questionnaire.

INTERVENTIONS:
Other: A short, animated storytelling video on dietary sodium — Participants in the Intervention Arm will view a short, animated storytelling video on dietary sodium and the risks of cardiovascular disease due to increased intake of sodium.
  Arms: Intervention Arm
Other: A short, animated storytelling attention placebo video — The Attention Placebo Control Arm will view an attention placebo control video, unrelated to the outcomes measured in this trial.
  Arms: Attention Placebo Control Arm

SUMMARY:
This study will evaluate the effect of a short, animated storytelling intervention video on sodium intake as a major risk factor for cardiovascular disease on immediate and medium-term retention of knowledge about the risks of cardiovascular diesaes due to increased sodium intake. We will also measure voluntary engagement with the content of the short, animated storytelling intervention video on positive psychological capital.

In this 4-armed, parallel, randomized controlled trial, 10,000 adult, US participants will be randomly assigned to (1) a short, animated storytelling intervention video on sodium as a cardiovascular disease risk factor followed by surveys assessing the facts om sodium and cardiovascular disease conveyed in the video (2) the surveys only, (3) an attention placebo control video followed by the before mentioned surveys, and (4) an arm that is exposed to neither the video nor the surveys. Two weeks later, participants in all four arms will complete all of the surveys.

The primary outcome is knowledge about the cardiovascular disease risk associated with increased sodium intake (immediate and medium-term). The major scondary outcome is the extent of voluntary engagement with the short, animated storytelling video content.

ELIGIBILITY:
Inclusion Criteria:

* Registration with the Prolific Academic platform

Exclusion Criteria:

* none

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Immediate effect of the short, animated storytelling intervention video on knowledge about dietary sodium as a cardiovascular risk factor | immediately after watching the video
  The immediate effect of the short, animated storytelling intervention video on knowledge about dietary sodium as a cardiovascular risk factor assessed by a sodium questionnaire containing 30 questions.
Medium-term effect of the short, animated storytelling intervention video on knowledge about dietary sodium as a cardiovascular risk factor | 2 weeks after watching the video
  The medium-term effect of the short, animated storytelling intervention video on knowledge about dietary sodium as a cardiovascular risk factor assessed by a sodium questionnaire containing 30 questions.

SECONDARY OUTCOMES:
Immediate effect of the short, animated storytelling intervention video on behavioral expectation to reduce dietary sodium. | immediately after watching the video
  The immediate effect of the short, animated storytelling intervention video on behavioral expectation to reduce dietary sodium assessed by a questionnaire containing 30 questions on behavioral expectation.
Medium-term effect of the short, animated storytelling intervention video on behavioral expectation to reduce dietary sodium. | 2 weeks after watching the video
  The medium-term effect of the short, animated storytelling intervention video on behavioral expectation to reduce dietary sodium assessed by a questionnaire containing 30 questions on behavioral expectation.
Voluntary post-trial engagement (frequency) with the video content. | 2 weeks after entering the trial
  Assessment of the frequency (absolute number) of watching the trial videos after completion of the trial questionnaires
Voluntary post-trial engagement (duration) with the video content. | 2 weeks after entering the trial
  Assessment of the duration (in minutes) of watching the trial videos after completion of the trial questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Till Bärnighausen, Prof. Dr., Principal Investigator — Heidelberg University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adam M, Rohr JK, Greuel M, Nguyen VK, El Aziz MA, Uberreiter C, Coles O, Barnighausen T, Supady A. Digital storytelling boosts knowledge and behavioral expectation to reduce dietary sodium: a randomized controlled trial. NPJ Digit Med. 2026 Jan 9;9(1):21. doi: 10.1038/s41746-025-02258-x. PMID 41514069
- [Derived] Supady A, Nguyen K, Aziz MAE, Uberreiter C, Barnighausen T, Adam M. A short, animated storytelling video about sodium intake as a major cardiovascular risk factor and recommendations for a healthy diet: an online, randomized, controlled trial. Trials. 2023 Jun 10;24(1):390. doi: 10.1186/s13063-023-07418-6. PMID 37296468